CLINICAL TRIAL: NCT02655016
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Niraparib Maintenance Treatment in Patients With Advanced Ovarian Cancer Following Response on Front-Line Platinum-Based Chemotherapy
Brief Title: A Study of Niraparib (GSK3985771) Maintenance Treatment in Participants With Advanced Ovarian Cancer Following Response on Front-Line Platinum-Based Chemotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 213359; PR-30-5017-C (Other: Tesaro); 2023-508010-42 (Other: CTIS)
Record Dates: First submitted 2015-12-08; First posted 2016-01-13 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Cancer; Niraparib; GSK3985771; Poly(adenosine diphosphate [ADP]-ribose) polymerase (PARP)Inhibitor; Homologous recombination deficiency (HRD); HRD positive; PRIMA; PRIMA Clinical Trial; PRIMA Study
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Niraparib (Experimental)
  Interventions: Drug: Niraparib
- Participants receiving Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered.
  Arms: Participants receiving Niraparib
Drug: Placebo — Placebo will be administered.
  Arms: Participants receiving Placebo

SUMMARY:
This study aims to assess efficacy of Niraparib (GSK3985771) as maintenance treatment in participants with Stage III or IV ovarian cancer. Participants must have completed front-line platinum based regimen with complete response (CR) or partial response (PR). Data collection for Secondary Outcome measures is ongoing and the approximate duration of the study will be 7 years.

ELIGIBILITY:
Inclusion criteria:

* Participants must have histologically diagnosed high-grade serous or endometrioid, or high-grade predominantly serous or endometrioid ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that is Stage III or IV according to Federation Internationale de Gynécologie et d'Obstétrique (FIGO) criteria.
* Participants with inoperable Stage III and IV disease; All Stage IV participants with operable disease; Participants with stage III or IV disease treated with neoadjuvant chemotherapy and interval debulking surgery; and Participants with stage III disease who have visible residual disease after primary debulking surgery.
* Participants who have received intraperitoneal chemotherapy; All participants must have had more than or equal to (>=)6 and less than or equal to (<=)9 cycles of platinum-based therapy; Participants must have had >=2 post-operative cycles of platinum-based therapy following interval debulking surgery; Participants must have physician assessed Complete response (CR) or Partial response (PR) after >=3 cycles of therapy; and Participants must have either Cancer antigen 125 (CA-125) in the normal range or CA-125 decrease by more than 90 percent(%) during their front-line therapy that is stable for at least 7 days (no increase more than (>)15% from nadir).
* Participants must be randomized within 12 weeks of the first day of the last cycle of chemotherapy.
* All participants must agree to undergo central tumor HRD testing.
* Participants of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin [hCG]) within 7 days prior to receiving the first dose of study treatment.

Exclusion criteria:

* Participant has mucinous or clear cell subtypes of epithelial ovarian cancer, carcinosarcoma or undifferentiated ovarian cancer.
* Participants with Stage III disease who have had complete cytoreduction (no visible residual disease) after primary debulking surgery.
* Participant has undergone more than two debulking surgeries for the study disease.
* Participant is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for up to 180 days after the last dose of study treatment.
* Participant has a known hypersensitivity to the components of niraparib or its excipients.
* Participant has received prior treatment with a known PARP inhibitor or has participated in a study where any treatment arm included administration of a known PARP inhibitor.
* Participant is to receive bevacizumab as maintenance treatment.
* Participant has had investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Participant has had any known >=Grade 3 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted >4 weeks.
* Participant has a condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results or interfere with the participation for the full duration of the study treatment, including:

  1. Participant received a transfusion (platelets or red blood cells) within 2 weeks of the first dose of study treatment.
  2. Participant received colony-stimulating factors (e.g., granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study treatment.
* Participant has been diagnosed and/or treated for invasive cancer less than 5 years prior to study enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 733 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (104):
- United States (44):
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Geneva, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Harrison, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Kennewick, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Belgium (7):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Libramont
  - GSK Investigational Site, Namur
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Odense C
- Finland (4):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- GSK Investigational Site, Angers, France
- Germany (9):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Fürth
  - GSK Investigational Site, Göttingen
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Hildesheim
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Dunmore RoadWaterford
  - GSK Investigational Site, Galway
- Israel (3):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
- Italy (4):
  - GSK Investigational Site, Lecce
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Napoli
- GSK Investigational Site, Oslo, Norway
- Spain (10):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Sweden (2):
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Switzerland (4):
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Frauenfeld
  - GSK Investigational Site, Zurich
- United Kingdom (8):
  - GSK Investigational Site, Blackburn
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monk BJ, Barretina-Ginesta MP, Pothuri B, Vergote I, Graybill W, Mirza MR, McCormick CC, Lorusso D, Moore RG, Freyer G, O'Cearbhaill RE, Heitz F, O'Malley DM, Redondo A, Shahin MS, Vulsteke C, Bradley WH, Haslund CA, Chase DM, Pisano C, Holman LL, Perez MJR, DiSilvestro P, Gaba L, Herzog TJ, Bruchim I, Compton N, Shtessel L, Malinowska IA, Gonzalez-Martin A. Niraparib first-line maintenance therapy in patients with newly diagnosed advanced ovarian cancer: final overall survival results from the PRIMA/ENGOT-OV26/GOG-3012 trial. Ann Oncol. 2024 Nov;35(11):981-992. doi: 10.1016/j.annonc.2024.08.2241. Epub 2024 Sep 14. PMID 39284381
- [Derived] Monk BJ, Romero I, Graybill W, Churruca C, O'Malley DM, Knudsen AO, Yap OWS, Baurain JF, Rose PG, Denys H, Ghamande S, Pisano C, Fabbro M, Braicu EI, Calvert PM, Amit A, Prendergast E, Taylor A, Kheibarshekan L, Zhang ZY, Zajic S, Jewell RC, Gupta D, Gonzalez-Martin A. Niraparib Population Pharmacokinetics and Exposure-Response Relationships in Patients With Newly Diagnosed Advanced Ovarian Cancer. Clin Ther. 2024 Aug;46(8):612-621. doi: 10.1016/j.clinthera.2024.06.001. Epub 2024 Jul 16. PMID 39019698
- [Derived] Vulsteke C, Chambers SK, Perez MJR, Chan JK, Raaschou-Jensen N, Zhuo Y, Lorusso D, Herzog TJ, de la Motte Rouge T, Thomes Pepin JA, Braicu EI, Chen LM, Levy T, Barter JF, Pilar Barretina-Ginesta M, Joosens E, York W, Malinowska IA, Gonzalez-Martin A, Monk BJ. Tolerability of the niraparib individualized starting dose in the PRIMA/ENGOT-OV26/GOG-3012 trial of niraparib first-line maintenance therapy. Eur J Cancer. 2024 Sep;208:114157. doi: 10.1016/j.ejca.2024.114157. Epub 2024 Jun 10. PMID 39013265
- [Derived] Graybill WS, Pardo Burdalo B, O'Malley DM, Vergote I, Monk BJ, Auranen A, Copeland LJ, Sabbatini R, Herzog TJ, Follana P, Pothuri B, Braicu EI, McCormick C, Yubero A, Moore RG, Vuylsteke P, Raaschou-Jensen N, York W, Hartman J, Gonzalez-Martin A. Predictors of long-term progression-free survival in patients with ovarian cancer treated with niraparib in the PRIMA/ENGOT-OV26/GOG-3012 study. Int J Gynecol Cancer. 2024 Jul 1;34(7):1041-1050. doi: 10.1136/ijgc-2024-005356. PMID 38950925
- [Derived] Valabrega G, Pothuri B, Oaknin A, Graybill WS, Sanchez AB, McCormick C, Baurain JF, Tinker AV, Denys H, O'Cearbhaill RE, Hietanen S, Moore RG, Knudsen AO, de La Motte Rouge T, Heitz F, Levy T, York W, Gupta D, Monk BJ, Gonzalez-Martin A. Efficacy and safety of niraparib in patients aged 65 years and older with advanced ovarian cancer: Results from the PRIMA/ENGOT-OV26/GOG-3012 trial. Gynecol Oncol. 2024 Aug;187:128-138. doi: 10.1016/j.ygyno.2024.03.009. Epub 2024 Jun 3. PMID 38833992
- [Derived] Gonzalez-Martin A, Pothuri B, Vergote I, Graybill W, Lorusso D, McCormick CC, Freyer G, Backes F, Heitz F, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Malinowska IA, Shtessel L, Compton N, Mirza MR, Monk BJ. Progression-free survival and safety at 3.5 years of follow-up: results from the randomized phase 3 PRIMA/ENGOT-OV26/GOG-3012 trial of niraparib maintenance treatment in patients with newly diagnosed ovarian cancer - a plain language summary. Future Oncol. 2024;20(22):1531-1544. doi: 10.2217/fon-2023-0782. Epub 2024 Mar 19. PMID 38501262
- [Derived] Pothuri B, Han S, Chase DM, Heitz F, Burger RA, Gaba L, Van Le L, Guerra E, Bender D, Korach J, Cloven N, Churruca C, Follana P, DiSilvestro P, Baurain JF, Jardon K, Pisano C, Peen U, Maenpaa J, Gupta D, Bacque E, Li Y, Compton N, Antonova J, Monk BJ, Gonzalez-Martin A. Health-related quality of life in patients with newly diagnosed advanced ovarian cancer treated with niraparib vs placebo: Results from the phase 3 randomized PRIMA/ENGOT-OV26/GOG-3012 trial. Gynecol Oncol. 2024 May;184:168-177. doi: 10.1016/j.ygyno.2024.01.021. Epub 2024 Feb 6. PMID 38325276
- [Derived] Gonzalez-Martin A, Pothuri B, Vergote I, Graybill W, Lorusso D, McCormick CC, Freyer G, Backes F, Heitz F, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Malinowska IA, Shtessel L, Compton N, Mirza MR, Monk BJ. Progression-free survival and safety at 3.5years of follow-up: results from the randomised phase 3 PRIMA/ENGOT-OV26/GOG-3012 trial of niraparib maintenance treatment in patients with newly diagnosed ovarian cancer. Eur J Cancer. 2023 Aug;189:112908. doi: 10.1016/j.ejca.2023.04.024. Epub 2023 May 3. PMID 37263896
- [Derived] Barretina-Ginesta MP, Monk BJ, Han S, Pothuri B, Auranen A, Chase DM, Lorusso D, Anderson C, Abadie-Lacourtoisie S, Cloven N, Braicu EI, Amit A, Redondo A, Shah R, Kebede N, Hawkes C, Gupta D, Woodward T, O'Malley DM, Gonzalez-Martin A. Quality-adjusted time without symptoms of disease or toxicity and quality-adjusted progression-free survival with niraparib maintenance in first-line ovarian cancer in the PRIMA trial. Ther Adv Med Oncol. 2022 Sep 22;14:17588359221126149. doi: 10.1177/17588359221126149. eCollection 2022. PMID 36172173
- [Derived] O'Cearbhaill RE, Perez-Fidalgo JA, Monk BJ, Tusquets I, McCormick C, Fuentes J, Moore RG, Vulsteke C, Shahin MS, Forget F, Bradley WH, Hietanen S, O'Malley DM, Dorum A, Slomovitz BM, Baumann K, Selle F, Calvert PM, Artioli G, Levy T, Kumar A, Malinowska IA, Li Y, Gupta D, Gonzalez-Martin A. Efficacy of niraparib by time of surgery and postoperative residual disease status: A post hoc analysis of patients in the PRIMA/ENGOT-OV26/GOG-3012 study. Gynecol Oncol. 2022 Jul;166(1):36-43. doi: 10.1016/j.ygyno.2022.04.012. Epub 2022 May 9. PMID 35550709
- [Derived] Gonzalez-Martin A, Pothuri B, Vergote I, DePont Christensen R, Graybill W, Mirza MR, McCormick C, Lorusso D, Hoskins P, Freyer G, Baumann K, Jardon K, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Lund B, Backes F, Barretina-Ginesta P, Haggerty AF, Rubio-Perez MJ, Shahin MS, Mangili G, Bradley WH, Bruchim I, Sun K, Malinowska IA, Li Y, Gupta D, Monk BJ; PRIMA/ENGOT-OV26/GOG-3012 Investigators. Niraparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2391-2402. doi: 10.1056/NEJMoa1910962. Epub 2019 Sep 28. PMID 31562799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this double-blind, randomized, placebo-controlled study, participants with stage III or IV ovarian cancer were randomized to receive either niraparib or placebo in 2:1 ratio. The results presented are based on the primary analysis up to month 34. Data collection is still on-going and additional results will be provided after study completion (7 years).
Pre-assignment Details: A total of 989 participants were screened, of which 256 participants did not meet eligibility criteria. A total of 733 participants were enrolled and randomized in the study, of which 728 participants received study treatment (4 participants were screen failures after randomization and 1 participant withdrew consent before first dose).
Groups:
- Placebo: Participants received placebo matching niraparib 300 milligram (mg) (3×100 mg capsules) (fixed dose) once daily (QD) orally beginning on Day 1 of every cycle (each cycle of 28-days) in a double-blind fashion until a modified starting dose regimen was implemented in protocol amendment. After the protocol amendment, participants received placebo based upon the participant's Baseline body weight or Baseline platelet count (individualized dose): 300 mg (3×100 mg capsules for participants with a Baseline body weight >=77 kilogram [kg] and Baseline platelet count >=150,000 per microliter [μL]) or 200 mg (2×100 mg capsules for participants with a Baseline body weight <77 kg or Baseline platelet count <150,000 per μL).
- Niraparib: Participants received niraparib 300 mg (3×100 mg capsules) (fixed dose) QD orally beginning on Day 1 of every cycle (each cycle of 28-days) in a double-blind fashion until a modified starting dose regimen was implemented in protocol amendment. After the protocol amendment, participants received niraparib based upon the participant's Baseline body weight or Baseline platelet count (individualized dose): 300 mg (3×100 mg capsules for participants with a Baseline body weight >=77 kg and Baseline platelet count >=150,000 per μL) or 200 mg (2×100 mg capsules for participants with a Baseline body weight <77 kg or Baseline platelet count <150,000 per μL).
Period: Overall Study
Arm/Group | Placebo | Niraparib
Started | 246 | 487
Received Study Treatment | 244 (2 participants never received treatment due to screen failure after randomization.) | 484 (3 participants never received treatment (2 failed screening & 1 withdrew consent before first dose).)
Ongoing With Treatment in the Study | 69 | 177
Completed | 191 (69 participants are ongoing in the study.) | 397 (177 participants are ongoing in the study.)
Not Completed | 55 | 90
Not completed — Disease progression | 6 | 4
Not completed — Site closed | 0 | 1
Not completed — Death | 30 | 48
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 18 | 36

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for all randomized participants including 5 randomized participants who never received treatment (4-Screen failure and 1-Withdrew consent).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Niraparib | Total
Number analyzed (Participants) | 246 | 487 | 733
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (10.39) | 61.1 (10.79) | 61.2 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 487 | 733
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 219 | 436 | 655
  Black | 2 | 10 | 12
  Asian | 11 | 14 | 25
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Unknown | 14 | 25 | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from the date of treatment randomization to the date of first documentation of disease progression or death due to any cause in the absence of documented progression, whichever occurs first. It was assessed by the blinded independent central review (BICR). Median and 95% confidence interval (CI) are presented.
Time Frame: Up to 34 months
Population: Intent-to-Treat (ITT) population comprised of all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 246 | 487
Months | 8.2 [7.3 to 8.5] | 13.8 [11.5 to 14.9]
Statistical Analysis 1: Comparison: Placebo vs Niraparib; Test type: Superiority; p < 0.0001, Log Rank — p-value was calculated based on stratified log-rank test using randomization stratification factors: administration of neoadjuvant chemotherapy, best response to platinum therapy and homologous recombination deficiency (HRD) status; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.502 to 0.755] — If hazard ratio was found to be <1 then niraparib can be considered as superior to placebo

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death by any cause. Median and 95% CI are presented for overall survival interim analysis.
Time Frame: Up to 34 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 246 | 487
Months | NA [25.0 to NA] — NA indicates median and 95% CI (upper limit) could not be derived, as <50% of participants experienced the event within the treatment arm. | 30.3 [30.3 to NA] — NA indicates 95% CI (upper limit) could not be derived, as <75% of participants experienced the event within the treatment arm.
Statistical Analysis 1: Comparison: Placebo vs Niraparib; Test type: Superiority; p = 0.1238, Log Rank — p-value was calculated based on stratified log-rank test using randomization stratification factors: administration of neoadjuvant chemotherapy, best response to platinum therapy and HRD status; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.442 to 1.106] — If hazard ratio was found to be <1 then niraparib can be considered as superior to placebo

3. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: Time to first subsequent therapy was defined as the time from the date of randomization to the date of the first subsequent anti-cancer therapy or death, whichever occurs first. Median and 95% CI are presented.
Time Frame: Up to 34 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 246 | 487
Months | 12.0 [10.3 to 13.9] | 18.6 [15.8 to 24.7]
Statistical Analysis 1: Comparison: Placebo vs Niraparib; Test type: Superiority; p = 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.521 to 0.802] — If hazard ratio was found to be <1 then niraparib can be considered as superior to placebo

4. Secondary Outcome: Progression-Free Survival-2 (PFS2)
Description: PFS2 was defined as the time from the date of randomization to the date of progression on the next anti-cancer therapy following study treatment or death by any cause, whichever occurs first. Median and 95% CI are presented.
Time Frame: Up to 34 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 246 | 487
Months | NA [NA to NA] — NA indicates median and 95% CI could not be derived, as <25% of participants experienced the event within the treatment arm. | 27.2 [25.3 to NA] — NA indicates 95% CI (upper limit) could not be derived, as <75% of participants experienced the event within the treatment arm.
Statistical Analysis 1: Comparison: Placebo vs Niraparib; Test type: Superiority; p = 0.2242, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.577 to 1.139] — If hazard ratio was found to be <1 then niraparib can be considered as superior to placebo

5. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO): Functional Assessment of Cancer Therapy-Ovarian Symptom Index (FOSI)
Description: FOSI is a validated, 8-item measure of symptom response to treatment for ovarian cancer. Participants responded to their symptom experience over the past 7 days using a 5-point Likert scale scored from "not at all" (0) to "very much" (4). FOSI score was calculated as (sum of item scores)*8 divided by (number of items answered). The FOSI score ranged from 0 (severely symptomatic) to 32 (asymptomatic). A higher score indicated a better quality of life (QoL). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 240 | 479
Scores on a scale | -0.3 (0.22) | -0.4 (0.15)

6. Secondary Outcome: Change From Baseline in PRO: European Quality of Life Scale, 5-dimensions, 5-levels of Severity (EQ-5D-5L) Utility Score
Description: The EQ-5D-5L is a well-validated general preference-based, health-related QoL instrument. The five-item measure has 1 question assessing each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 243 | 477
Scores on a scale | 0.005 (0.0066) | 0.016 (0.0046)

7. Secondary Outcome: Change From Baseline in Functional Scales of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC-QLQ-C30)
Description: EORTC-QLQ-C30 incorporates 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), a global health status/QoL scale (global health status, QoL), and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulty) assessing additional symptoms commonly reported by participants with cancer. Five functional scales had total 15 items (physical-5, role-2, cognitive-4, emotional-2, and social-2). Each functional scales score was calculated by averaging scores of all scale items and transforming average scores linearly (1 minus [average score minus 1] divided by 3*100). All of the functional scales range in score from 0 to 100. Higher score represents a higher ("better") level of functioning. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 244 | 479
Scores on a scale
  Physical Functioning, n=244,479 | 2.119 (0.8131) | 2.013 (0.5735)
  Role Functioning, n=244,479 | 2.341 (1.2427) | 1.590 (0.8810)
  Emotional Functioning, n=243,478: number analyzed (Participants) | 243 | 478
  Emotional Functioning, n=243,478 | -0.011 (1.1218) | -0.870 (0.7685)
  Cognitive Functioning, n=243,478: number analyzed (Participants) | 243 | 478
  Cognitive Functioning, n=243,478 | -0.020 (1.2105) | -0.842 (0.7952)
  Social Functioning, n=243,478: number analyzed (Participants) | 243 | 478
  Social Functioning, n=243,478 | 5.557 (1.2449) | 4.445 (0.8633)

8. Secondary Outcome: Change From Baseline in Global Health Status/QoL of EORTC-QLQ-C30
Description: EORTC-QLQ-C30 incorporates 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), a global health status/QoL scale (global health status, QoL), and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulty) assessing additional symptoms commonly reported by participants with cancer. A global health status/QoL scale had total 2 items. Each global health status/QoL scales score was calculated by averaging scores of all scale items and transforming average scores linearly ([average score minus 1] divided by 6*100). The global health status/QoL scales range in score from 0 to 100. Higher score represents a higher ("better") level of health status/QoL. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 243 | 478
Scores on a scale | 1.177 (1.0005) | 1.009 (0.6898)

9. Secondary Outcome: Change From Baseline in Symptoms Scales and Symptoms Items (Dyspnea, Appetite Loss, Insomnia, Constipation, Diarrhea and Financial Difficulty) of EORTC-QLQ-C30
Description: EORTC-QLQ-C30 incorporates 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), a global health status/QoL scale, and 6 single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulty) assessing additional symptoms commonly reported by participants with cancer. Symptom scale had total 7 items (fatigue-3, pain-2, nausea/vomiting-2). Each symptoms scales and 6 single additional symptoms items score was calculated by averaging scores of all scale items and transforming average scores linearly ([average score minus 1] divided by 3*100). All of the symptoms scales and 6 single additional symptoms scales range in score from 0 to 100. Higher score represents a higher ("worse") level of symptoms. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 244 | 480
Scores on a scale
  Fatigue, n=243,479: number analyzed (Participants) | 243 | 479
  Fatigue, n=243,479 | -0.082 (1.2394) | 0.085 (0.8363)
  Nausea/Vomiting, n=244,479: number analyzed (Participants) | 244 | 479
  Nausea/Vomiting, n=244,479 | 1.673 (0.7595) | 3.115 (0.4828)
  Pain, n=244,480 | -0.195 (1.2274) | 0.765 (1.0166)
  Dyspnea, n=244,479: number analyzed (Participants) | 244 | 479
  Dyspnea, n=244,479 | 0.644 (1.3592) | 1.347 (0.8518)
  Insomnia, n=244,479: number analyzed (Participants) | 244 | 479
  Insomnia, n=244,479 | 2.195 (1.9882) | 3.478 (1.2791)
  Appetite Loss, n=8,30: number analyzed (Participants) | 8 | 30
  Appetite Loss, n=8,30 | -0.827 (4.3987) | -0.395 (2.3195)
  Constipation, n=244,478: number analyzed (Participants) | 244 | 478
  Constipation, n=244,478 | -1.147 (1.5793) | 6.356 (1.0446)
  Diarrhea, n=8,30: number analyzed (Participants) | 8 | 30
  Diarrhea, n=8,30 | 9.335 (3.8667) | -3.340 (2.0136)
  Financial Difficulties, n=243,475: number analyzed (Participants) | 243 | 475
  Financial Difficulties, n=243,475 | -5.058 (1.2978) | -3.356 (0.9276)

10. Secondary Outcome: Change From Baseline in Functional Scales of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Ovarian Cancer Module (EORTC-QLQ-OV28)
Description: EORTC-QLQ-OV28 is supplement to EORTC-QLQ-C30. It includes 3 functional scales (body image, sexuality, attitude to disease/treatment) and 5 symptom scales/items (abdominal/gastrointestinal [GI] symptoms, peripheral neuropathy, hormonal/menopausal symptoms, other chemotherapy side-effects, and hair loss). Functional scales score (body Image and attitude to disease/treatment) was calculated by averaging scores of all scale items and transforming average scores linearly (1 minus [average score minus 1] divided by 3*100). Functional scales score (sexuality) was calculated by averaging scores of all scale items and transforming average scores linearly ([average score minus 1] divided by 3*100). All of the functional scales range in score from 0 to 100. Higher score represents a higher ("better") level of functioning. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to 34 months
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 244 | 475
Scores on a scale
  Body Image, n=244,475 | 10.069 (1.4820) | 8.488 (1.0138)
  Sexuality, n=240,471: number analyzed (Participants) | 240 | 471
  Sexuality, n=240,471 | 3.257 (1.1886) | 3.625 (0.8004)
  Attitude to disease/Treatment, n=244,475 | 12.216 (1.3257) | 13.660 (0.9309)

11. Secondary Outcome: Change From Baseline in Symptoms Scale of EORTC-QLQ-OV28
Description: EORTC-QLQ-OV28 is supplement to EORTC-QLQ-C30. It includes 3 functional scales (body image, sexuality, attitude to disease/treatment) and 5 symptom scales/items (abdominal/GI symptoms, peripheral neuropathy, hormonal/menopausal symptoms, other chemotherapy side-effects, and hair loss). Symptoms scales score was calculated by averaging scores of all scale items and transforming average scores linearly ([average score minus 1] divided by 3*100). All of the symptoms scales range in score from 0 to 100. Higher score represents a higher ("worse") level of symptoms. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose).
Time Frame: Baseline (Day 1, Pre-dose) and Up to 34 months
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 244 | 481
Scores on a scale
  Abdominal/GI, n=244,481 | 0.832 (0.8110) | 2.185 (0.5703)
  Peripheral Neuropathy, n=244,480: number analyzed (Participants) | 244 | 480
  Peripheral Neuropathy, n=244,480 | -9.629 (1.3219) | -8.217 (0.9295)
  Hormonal/Menopausal Symptoms, n=244,480: number analyzed (Participants) | 244 | 480
  Hormonal/Menopausal Symptoms, n=244,480 | -2.521 (1.3074) | 1.501 (0.8803)
  Other Chemotherapy Side Effects, n=244,480: number analyzed (Participants) | 244 | 480
  Other Chemotherapy Side Effects, n=244,480 | -3.023 (0.8358) | -2.219 (0.5581)
  Hair Loss, n=242,477: number analyzed (Participants) | 242 | 477
  Hair Loss, n=242,477 | -20.743 (1.3690) | -23.363 (0.9821)

12. Other Pre Specified Outcome: Number of Participants With Any Non-serious Adverse Event (Non-SAE) or Any SAE
Description: An adverse event is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE.
Time Frame: Up to 34 months
Population: Safety Population comprised of all participants who received at least 1 dose of study drug. 5 participants (2 participants from Placebo group and 3 participants from Niraparib group) out of 733 participants did not receive any study treatment and thus, were excluded from the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 244 | 484
Participants
  Any non-SAE | 223 | 478
  Any SAE | 32 | 156

13. Other Pre Specified Outcome: Area Under the Curve (AUC) From 0 to the Last Quantifiable Concentration (AUC[0-last])
Description: Blood samples were planned to be collected for assessment of AUC(0-last).
Time Frame: Up to 34 months
Population: ITT Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax)
Description: Blood samples were planned to be collected for assessment of Cmax.
Time Frame: Up to 34 months
Population: ITT Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Niraparib
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Number of Participants With Positive HRD Test
Description: Number of participants with positive HRD test was planned to be assessed.
Time Frame: Up to 34 months
Population: ITT Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Placebo | Niraparib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were reported from start of study treatment (Day 1) and up to month 34 (primary analysis)
Description: Non-SAEs and SAEs were presented for Safety Population. 5 participants out of 733 participants did not receive any study treatment and were excluded from the Safety Population. The results presented are based on the primary analysis up to month 34. Data collection is still on-going and additional results will be provided after study completion (7 years).
Arm/Group | Placebo | Niraparib
All-Cause Mortality (participants affected / at risk) | 31/244 | 48/484
Serious Adverse Events (participants affected / at risk) | 32/244 | 156/484
Other Adverse Events (participants affected / at risk) | 223/244 | 478/484
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=244) | Niraparib (N=484)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 27 (28)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 59 (65)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal fat apron (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 5 (6)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 14 (19)
Subileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (4) | 8 (10)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 20 (25)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (2)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fasting (Social circumstances) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=244) | Niraparib (N=484)
Anaemia (Blood and lymphatic system disorders) | 43 (83) | 306 (921)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 13 (27) | 57 (145)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 12 (40)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 16 (32) | 126 (366)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 210 (549)
Angina pectoris (Cardiac disorders) | 0 (0) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Metabolic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 5 (6) | 39 (45)
Sinus tachycardia (Cardiac disorders) | 3 (5) | 12 (17)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 6 (6) | 25 (28)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 6 (6)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Paraesthesia ear (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 4 (6) | 11 (11)
Vertigo (Ear and labyrinth disorders) | 6 (7) | 13 (13)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (2)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 2 (3)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 11 (12)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 4 (5)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid sensory disorder (Eye disorders) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (2)
Myopia (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (5)
Photophobia (Eye disorders) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Retinal exudates (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 5 (5)
Visual acuity reduced (Eye disorders) | 1 (1) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 5 (5)
Vitreous floaters (Eye disorders) | 0 (0) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 11 (11) | 15 (19)
Abdominal distension (Gastrointestinal disorders) | 30 (36) | 32 (36)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 4 (5)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 74 (102) | 105 (146)
Abdominal pain lower (Gastrointestinal disorders) | 13 (17) | 15 (16)
Abdominal pain upper (Gastrointestinal disorders) | 21 (26) | 41 (59)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 4 (6)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 2 (3) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 5 (5)
Ascites (Gastrointestinal disorders) | 8 (8) | 3 (3)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 46 (52) | 189 (262)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (2) | 2 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 55 (82) | 91 (132)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (8) | 40 (46)
Dyspepsia (Gastrointestinal disorders) | 14 (16) | 34 (43)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 6 (10)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Eructation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 2 (3)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 2 (3)
Flatulence (Gastrointestinal disorders) | 7 (12) | 17 (20)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 25 (28)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 3 (5) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 5 (6)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 3 (3)
Melaena (Gastrointestinal disorders) | 0 (0) | 4 (4)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 67 (100) | 278 (448)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral contusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 2 (3)
Oral mucosal discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3) | 7 (9)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (7)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (7) | 16 (18)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 6 (6)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 28 (34) | 108 (153)
Adhesion (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 31 (47) | 78 (138)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 3 (3)
Catheter site rash (General disorders) | 0 (0) | 1 (1)
Catheter site vesicles (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 5 (5)
Chest pain (General disorders) | 4 (4) | 3 (4)
Chills (General disorders) | 3 (3) | 6 (7)
Cyst (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 3 (4)
Early satiety (General disorders) | 2 (2) | 4 (4)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 72 (101) | 168 (242)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 3 (3)
Hernia pain (General disorders) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 11 (12) | 15 (22)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 7 (7)
Mass (General disorders) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 6 (10) | 23 (29)
Non-cardiac chest pain (General disorders) | 2 (2) | 13 (15)
Oedema peripheral (General disorders) | 11 (19) | 30 (35)
Pain (General disorders) | 6 (6) | 16 (17)
Peripheral swelling (General disorders) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 15 (17) | 41 (47)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 2 (8)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 2 (2) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Seasonal allergy (Immune system disorders) | 5 (5) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 12 (13)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 5 (7)
Cystitis (Infections and infestations) | 4 (4) | 6 (6)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 4 (4)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 4 (5) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 3 (3)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 1 (3) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 5 (8)
Hordeolum (Infections and infestations) | 0 (0) | 4 (4)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 6 (6)
Laryngitis (Infections and infestations) | 1 (2) | 2 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 4 (4)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 3 (4) | 7 (10)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (6)
Pneumonia (Infections and infestations) | 2 (2) | 8 (9)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 9 (10)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 7 (7) | 15 (27)
Skin candida (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 7 (9)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 18 (22) | 28 (31)
Urinary tract infection (Infections and infestations) | 19 (25) | 44 (48)
Vaginal infection (Infections and infestations) | 2 (2) | 3 (4)
Viral infection (Infections and infestations) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 25 (40) | 49 (55)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (5) | 22 (29)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 12 (14)
Foot fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mallet finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 6 (6)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (21) | 42 (67)
Amylase increased (Investigations) | 0 (0) | 3 (4)
Aspartate aminotransferase (Investigations) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 10 (16) | 43 (78)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 6 (8) | 42 (66)
Blood bilirubin increased (Investigations) | 0 (0) | 7 (13)
Blood calcium increased (Investigations) | 0 (0) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 4 (4)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 10 (12) | 55 (96)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 4 (6)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 3 (3)
Blood magnesium decreased (Investigations) | 0 (0) | 3 (4)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 5 (5)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (3) | 4 (4)
Bone density decreased (Investigations) | 1 (1) | 0 (0)
Carbohydrate antigen 125 increased (Investigations) | 10 (11) | 7 (7)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Eosinophil count decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 11 (21)
Haematocrit decreased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 5 (7)
Heart rate increased (Investigations) | 0 (0) | 9 (10)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (4) | 25 (43)
Mean cell volume increased (Investigations) | 0 (0) | 3 (4)
Monocyte count decreased (Investigations) | 0 (0) | 2 (2)
Monocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (10) | 82 (207)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 129 (338)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 3 (3)
Red blood cell count decreased (Investigations) | 0 (0) | 4 (4)
Sputum abnormal (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (6) | 20 (27)
Weight increased (Investigations) | 19 (30) | 17 (24)
White blood cell count decreased (Investigations) | 8 (16) | 74 (205)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (21) | 92 (112)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 6 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 9 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (8) | 19 (28)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (10)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (6) | 8 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 25 (37)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (18) | 38 (58)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 19 (35)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (10)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (77) | 85 (116)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (6)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (29) | 64 (84)
Bone disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (8)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4 (7) | 4 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (25) | 19 (24)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (15)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 12 (17)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 12 (15)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (4) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (18) | 36 (49)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 12 (13)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (10)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 14 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (20) | 38 (53)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Aura (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 6 (6)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 3 (5) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 26 (30) | 71 (96)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 10 (13) | 25 (34)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 36 (46) | 126 (190)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 8 (12)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (5) | 7 (7)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 3 (4) | 4 (5)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 15 (18) | 31 (38)
Neurotoxicity (Nervous system disorders) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 8 (9) | 11 (20)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (10) | 18 (21)
Polyneuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 3 (3) | 2 (3)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 4 (4)
Sciatica (Nervous system disorders) | 3 (4) | 9 (10)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 5 (6)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 7 (9)
Agitation (Psychiatric disorders) | 1 (1) | 8 (11)
Anxiety (Psychiatric disorders) | 19 (24) | 43 (53)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3)
Depressed mood (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 10 (14) | 26 (28)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 3 (3)
Genito-pelvic pain/penetration disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination, olfactory (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 35 (37) | 119 (162)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 3 (3)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1) | 3 (4)
Stress (Psychiatric disorders) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 4 (4)
Bladder pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 2 (2)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 10 (11) | 21 (22)
Haematuria (Renal and urinary disorders) | 6 (6) | 5 (6)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 2 (3)
Micturition urgency (Renal and urinary disorders) | 4 (4) | 3 (3)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 5 (5) | 11 (11)
Polyuria (Renal and urinary disorders) | 1 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 4 (4)
Urine odour abnormal (Renal and urinary disorders) | 1 (2) | 2 (2)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Breast calcifications (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 2 (4)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital paraesthesia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 6 (7) | 8 (8)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | 4 (6)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Vaginal mucosal blistering (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vulvovaginal dryness (Reproductive system and breast disorders) | 6 (6) | 7 (12)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 3 (4)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (45) | 74 (92)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 88 (129)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 17 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 23 (24)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 21 (28)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 22 (24)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 14 (16)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (12) | 19 (21)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (9)
Erythema dyschromicum perstans (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 28 (29)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 29 (35)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (21) | 13 (18)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 8 (12) | 23 (29)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (14)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Astringent therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (3) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 7 (7)
Hot flush (Vascular disorders) | 20 (20) | 54 (64)
Hyperaemia (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 17 (28) | 81 (142)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 3 (3)
Pallor (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT02655016/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02655016/SAP_001.pdf